CLINICAL TRIAL: NCT03845478
Title: Effect of the Prescription of 10,000 Steps a Day Using a Pedometer Via Mobile APP, Through a Goal Setting System, in the Body Composition of Overweight Adults: a 6-Month Randomized Weight Loss and mHealth Trial.
Brief Title: Effect of the Prescription of 10,000 Steps Per Day Using a Pedometer APP in the Body Composition of Overweight Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad de Córdoba (Other)
Responsible Party: Principal Investigator, Alberto Hernández de los Reyes, Principal Investigator, Universidad de Córdoba
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: A284R4156
Record Dates: First submitted 2019-02-15; First posted 2019-02-19 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Overweight; Obesity
Keywords: Obesity; Physical Activity; Fat mass; Fat free mass; Pedometer; mHealth
MeSH Terms: conditions — Overweight; Obesity; Motor Activity | interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (CG) (Active Comparator): Education, modifying diet and physical activity
  Interventions: Behavioral: Control Group (CG)
- Intervention Group (IG) (Experimental): Education and modifying diet and physical activity with prescription and goal setting
  Interventions: Behavioral: Intervention Group (IG)

INTERVENTIONS:
Behavioral: Control Group (CG) — The control group is subjected to follow a hypocaloric diet and receives information about the benefits of achieving 10,000 steps a day in weight loss and improved body composition.
  Arms: Control Group (CG)
Behavioral: Intervention Group (IG) — This group in addition to fulfilling a hypocaloric diet identical to the control group, and receive identical information about physical activity that the control group, it has a system of prescription, monitoring and establishing an objective to achieve 10,000 steps a day.
  Arms: Intervention Group (IG)

SUMMARY:
This study aimed the effect of the Accupedo pedometer smartphone app intervention, with goal setting of walking prescription of 10,000 steps per day, in overweight adults.

DETAILED DESCRIPTION:
The promotion of the increase in (FA) should be a priority in the treatment of weight loss in overweight or obese subjects. Walking is a solution to overcome physical inactivity, due to its low impact in which the person can control the intensity, duration and effort in order to reduce the risk of injury.

Monitoring the AF through the number of steps / day offers the possibility of standardizing the evaluation and monitoring. Although the goal of 10,000 steps a day may not be appropriate at various levels of age and physical condition, it is considered a reasonable and motivating goal for healthy adults and previous studies have demonstrated its effectiveness in weight loss programs.

The objective of this study is to compare the effect of the implementation of a monitoring system, goal to achieve, on physical activity in overweight and obese adults. Both groups, control and intervention, have a prescription of 10,000 steps a day to reach, but only the intervention group will have a control system, messages of encouragement and follow-up.

Participants (n=120) will be recruited through outpatient from private clinics in Cádiz, Andalucía, Spain, as well as through community presentations. Overweight or obese and sedentary adult will be randomly assigned into two groups.

For 6 months, all of the adults shall follow the same diet with an identical distribution of macronutrients. There will be a weekly check up of weight, fat, body water and muscle mass for all of them. The status of the number of steps in Accupedo is also checked every week

ELIGIBILITY:
Inclusion Criteria:

* Having a IMC >25,
* Being sedentary and
* Have not been submitted to a restrictive diet in the 6 months preceding this study.

Exclusion Criteria:

* Suffered from type 2 diabetes or renal conditions
* Being pregnancy or attempt at pregnancy,
* Being in a maternal lactation period,
* Being underage
* Undergoing antidepressant pharmacological treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 120 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline BMI | At baseline (0 years) and followed for 2 years
  Baseline mean BMI values will be measured and compared at 3, 6, 12 and 24 months. BMI will be assessed on a monthly basis during nutritional consultation through a Bioelectrical Impedance Analysis method using a Tanita BC-418 Segmental Body Composition Analyser/Scale
Changes from baseline Fatty mass | At baseline (0 years) and followed for 2 years
  Baseline mean Fatty mass values will be measured and compared at 3, 6, 12 and 24 months. Fatty mass will be assessed on a monthly basis during nutritional consultation through a Bioelectrical Impedance Analysis method using a Tanita BC-418 Segmental Body Composition Analyser/Scale. Fatty mass is measured as a percentage.
Changes from baseline Free-fatty mass | At baseline (0 years) and followed for 2 years
  Baseline mean Free-fatty mass values will be measured and compared at 3, 6, 12 and 24 months. Free-fatty mass will be assessed on a monthly basis during nutritional consultation through a Bioelectrical Impedance Analysis method using a Tanita BC-418 Segmental Body Composition Analyser/Scale. Fatty mass is measured as a percentage.
Changes from baseline Muscular Mass | At baseline (0 years) and followed for 2 years
  Baseline mean Muscular Mass values will be measured and compared at 3, 6, 12 and 24 months. Muscular Mass will be assessed on a monthly basis during nutritional consultation through a Bioelectrical Impedance Analysis method using a Tanita BC-418 Segmental Body Composition Analyser/Scale. Fatty mass is measured as a Kg.
Changes from baseline Corporal Water | At baseline (0 years) and followed for 2 years
  Baseline mean Corporal Water values will be measured and compared at 3, 6, 12 and 24 months. Corporal Water will be assessed on a monthly basis during nutritional consultation through a Bioelectrical Impedance Analysis method using a Tanita BC-418 Segmental Body Composition Analyser/Scale. Fatty mass is measured as a Kg.
Adherence to dietary pattern will be also measured through personal interview | At baseline (0 years) and followed for 2 years
  Participants will be subjected for an intervention based on nutritional (control group) and physical education (two intervention arms) during 24 months. Partial measures will be also taken every week. In the end of the trial, changes in dietary patterns will be measured comparing means differences between baselines, 3, 6, 12 and 24 months.
Adherence to physical activity patterns will be also measured through IPAQ (International Physical Activity Questionnaire) | At baseline (0 years) and followed for 2 years
  Participants will be subjected for an intervention based on nutritional (control group) and physical education (two intervention arms) during 24 months. Partial measures will be also taken every week. In the end of the trial, changes in physical activity will be measured comparing means differences between baselines, 3, 6, 12 and 24 months.
Changes from baseline in the number of steps per day | At baseline (0 years) and followed for 2 years
  Daily step-counts will be measured using Accupedo Pedometer app; this app can give feedback on distance, time and speed, and and average steps per day, week and month. Accupedo. Partial measures will be also taken every week. In the end of the trial, changes in physical activity patterns will be measured comparing means differences between baselines, 3, 6, 12 and 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Hernández-Reyes, Principal Investigator — Universidad de Córdoba

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hernandez-Reyes A, Camara-Martos F, Molina-Luque R, Moreno-Rojas R. Effect of an mHealth Intervention Using a Pedometer App With Full In-Person Counseling on Body Composition of Overweight Adults: Randomized Controlled Weight Loss Trial. JMIR Mhealth Uhealth. 2020 May 27;8(5):e16999. doi: 10.2196/16999. PMID 32348263